CLINICAL TRIAL: NCT02575820
Title: The Effects of Old Red Blood Cell Transfusion on Morbidity in Patients Undergoing Revision Total Hip Arthroplasty: Retrospective Study
Brief Title: Old Blood and Postoperative Complications
Status: Withdrawn | Type: Observational
Why Stopped: Sample size was too small to evaluate the clinical implications.
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Hyun-Jung Shin, Assistant Professor, Seoul National University Bundang Hospital
Other Study IDs: B-1510/318-112
Record Dates: First submitted 2015-10-11; First posted 2015-10-15 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2016-05

CONDITIONS: Orthopedics; Postoperative Complications; Red Blood Cells
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- RBC_old: shelf life of red blood cells of 15 or higher days
  Interventions: Procedure: Old red blood cells transfusion
- RBC_new: shelf life of red blood cells 14 or lower days
  Interventions: Procedure: New red blood cells transfusion

INTERVENTIONS:
Procedure: Old red blood cells transfusion — Red blood cells (shelf life > 14 days) transfusion during the operation (total hip replacement arthroplasty)
  Groups: RBC_old
Procedure: New red blood cells transfusion — Red blood cells (shelf life =< 14 days) transfusion during the operation (total hip replacement arthroplasty)
  Groups: RBC_new

SUMMARY:
The investigators sought to examine the effects of 'old' red blood cells on mortality and morbidity of patients who undergoing revision hip replacement arthroplasty. The investigators hypothesis is that patients have an increased risk of mortality and infection after 'old' red blood cells transfusions compared with those who received 'new' transfusions.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent revision total hip replacement

Exclusion Criteria:

* Patients who were not given red blood cells
* Patients who were given two units of which one unit was old and one was new

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent revision total hip replacement
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2015-11; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Mortality | postoperative 7 days
Sepsis | postoperative 7 days
Wound infection | postoperative 7 days
Postoperative delirium | postoperative 7 days
Postoperative bleeding | postoperative 7 days

SECONDARY OUTCOMES:
Transfusion related lung injury | postoperative 7 days
Pulmonary edema | postoperative 7 days
Pulmonary effusion | postoperative 7 days
Myocardial ischemia | postoperative 7 days
Pulmonary thromboembolism | postoperative 7 days
Renal failure | postoperative 7 days
Hepatic failure | postoperative 7 days

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, South Korea